CLINICAL TRIAL: NCT04355143
Title: Randomized, Open-Label, Controlled Trial of Colchicine to Reduce Cardiac Injury in Hospitalized COVID-19 (Coronavirus Disease 2019) Patients (COLHEART-19)
Brief Title: Colchicine to Reduce Cardiac Injury in COVID-19 (COLHEART-19)
Acronym: COLHEART-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-000685
Record Dates: First submitted 2020-04-14; First posted 2020-04-21 (Actual); Results first posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Random assignment to study arms in a 1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine plus current care (Experimental): Colchicine 0.6 mg po BID x 30 days plus current care per UCLA treating physicians
  Interventions: Drug: Colchicine Tablets; Other: Current care per UCLA treating physicians
- Current care alone (Active Comparator): Current care per UCLA physicians alone (control arm)
  Interventions: Other: Current care per UCLA treating physicians

INTERVENTIONS:
Drug: Colchicine Tablets — COLCRYS (colchicine, USP) tablets for oral administration, containing 0.6 mg of the active ingredient colchicine USP, administered po every 12 hours x 30 days.
  Other Names: COLCRYS; AR 374
  Arms: Colchicine plus current care
Other: Current care per UCLA treating physicians — Current care

SUMMARY:
Participants will be randomized in a 1:1 ratio to receive Colchicine plus current care per UCLA treating physicians versus current care per UCLA treating physicians alone (control arm). Importantly, this adaptive trial design allows for patients in either study arm to receive other investigational drugs for COVID-19 as new science emerges.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 infection by polymerase chain reaction
* Cardiac injury, including any of the following:

  * Elevated troponin level
  * Elevated B-type natriuretic peptide (BNP) level
  * New ischemic or arrhythmogenic changes on ECG/telemetry
  * New decrease in left ventricular ejection fraction (LVEF) or new pericardial effusion on echocardiogram
* Able to provide informed consent

Exclusion Criteria:

* Pregnancy, breastfeeding mothers, and women of childbearing age who are unable to use 2 forms of contraception, which includes:

  * Intrauterine devices (IUD), contraceptive implants, or tubal sterilization
  * Hormone methods with a barrier method
  * Two barrier methods
  * If a partner's vasectomy is the chosen method of contraception, a hormone or barrier method must also be used in conjunction
* Co-administration of Cytochrome P450 3A4 (CYPA3A4) and P-glycoprotein (P-gp) transport system inhibitors
* Concurrent use of strong CYP3A4 or P-gp inhibitors in patients with renal or hepatic impairment;
* Severe hematologic or neuromuscular disorders
* Severe renal impairment with concomitant hepatic impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Ardehali, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - UCLA Santa Monica Hospital, Santa Monica, California
  - Miami Cardiac and Vascular Institutde, Baptist Health South Florida, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rabbani A, Rafique A, Wang X, Campbell D, Wang D, Brownell N, Capdevilla K, Garabedian V, Chaparro S, Herrera R, Parikh RV, Ardehali R. Colchicine for the Treatment of Cardiac Injury in Hospitalized Patients With Coronavirus Disease-19. Front Cardiovasc Med. 2022 Jun 17;9:876718. doi: 10.3389/fcvm.2022.876718. eCollection 2022. PMID 35783822
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 304 screened individuals that met inclusion criteria,169 met exclusion criteria, 11 had co-enrollment conflicts with other clinical trials, 31 declined to participate.
Groups:
- Colchicine Plus Current Care: Colchicine 0.6 mg po BID (twice a day) x 30 days plus current care per UCLA treating physicians
  Colchicine Tablets: COLCRYS (colchicine, USP) tablets for oral administration, containing 0.6 mg of the active ingredient colchicine USP, administered po every 12 hours x 30 days.
  Current care per UCLA treating physicians: Current care
Period: Overall Study
Arm/Group | Colchicine Plus Current Care | Current Care Alone
Started | 48 | 45
Completed | 48 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colchicine Plus Current Care | Current Care Alone | Total
Number analyzed (Participants) | 48 | 45 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.2 (17) | 71.5 (19.5) | 71.3 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 21 | 30
  Male | 39 | 24 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28 | 21 | 49
  Black | 2 | 4 | 6
  Other | 18 | 20 | 38
Region of Enrollment [Number; unit: participants]
  United States | 48 | 45 | 93
Clinical Risk Factors [Count of Participants; unit: Participants]
  Hypertension | 39 | 34 | 73
  Hyperlipidemia | 35 | 23 | 58
  Diabetes | 19 | 16 | 35
  Tobacco use (current or former) | 14 | 19 | 33
  Cerebrovascular Disease | 4 | 8 | 12
  Chronic Kidney Disease | 18 | 8 | 26
  COPD | 5 | 5 | 10
  Other Lung Disease | 5 | 5 | 10
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index is an estimate of body fat based on body weight (kg) divided by height (m) squared. Population: Participants for whom BMI measurements were recorded at baseline.
  kg/m^2
    number analyzed (Participants) | 48 | 44 | 92
    (all) | 29.6 (6.9) | 28.4 (8.0) | 29.0 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Composite of All-cause Mortality, Need for Mechanical Ventilation, or Need for Mechanical Circulatory Support (MCS)
Description: Number of participants experiencing any of the following: All-cause mortality, need for mechanical ventilation, or need for mechanical circulatory support (MCS)
Time Frame: 90 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Plus Current Care | Current Care Alone
Number analyzed (Participants) | 48 | 45
Participants | 9 | 6

2. Secondary Outcome: Delta (Peak Minus Baseline) Troponin Level
Description: Change from initial troponin level to maximum level of troponin among measures taken during hospitalization and at 30 days
Time Frame: Baseline (Day 1), Day 30, Days 3 and 7 if hospitalized
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Colchicine Plus Current Care | Current Care Alone
Number analyzed (Participants) | 48 | 45
ng/mL
  Baseline | 0.1 (0.1) | 0.10 (0.5)
  Peak | 0.2 (0.4) | 0.1 (0.5)
  Delta | 0.1 (0.3) | 0 (0)

3. Secondary Outcome: Delta (Baseline to Peak) Brain Natriuretic Peptide (BNP) Level
Description: Change from baseline BNP level (Day 1) to maximum level of BNP among measures taken during hospitalization and at 30 days
Time Frame: Baseline (Day 1), Day 30, Days 3 and 7 if hospitalized
Population: Participants with analyzable samples at each timepoint
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Colchicine Plus Current Care | Current Care Alone
Number analyzed (Participants) | 48 | 45
pg/mL
  Baseline: number analyzed (Participants) | 48 | 43
  Baseline | 503 (765) | 389 (798)
  Peak: number analyzed (Participants) | 48 | 44
  Peak | 611 (796) | 514 (817)
  Delta: number analyzed (Participants) | 48 | 43
  Delta | 108 (218) | 134 (241)

4. Secondary Outcome: Change in Left Ventricular Ejection Fraction (LVEF) on Echocardiography
Description: Number of participants experiencing LVEF of < 50% on echocardiogram with failure to show an improvement of ≥ 5% at 30 days
Time Frame: Baseline, Day 30
Population: no participant was able to receive a repeat echocardiogram at day 30
Arm/Group | Colchicine Plus Current Care | Current Care Alone
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Delta (Peak Minus Baseline) C-Reactive Protein (CRP) Inflammatory Biomarker Level
Description: Change from baseline CRP level (Day 1) to maximum level of CRP among measures taken during hospitalization and at 30 days
Time Frame: Baseline (Day 1), Day 30, Days 3 and 7 if hospitalized
Population: Participants with analyzable samples at each timepoint
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Colchicine Plus Current Care | Current Care Alone
Number analyzed (Participants) | 48 | 45
mg/dL
  Baseline: number analyzed (Participants) | 47 | 45
  Baseline | 9.9 (7.3) | 7.2 (5.7)
  Peak | 13.6 (8.9) | 9.8 (7.8)
  Delta: number analyzed (Participants) | 47 | 45
  Delta | 3.9 (7.2) | 2.6 (4.1)

6. Secondary Outcome: Delta (Peak Minus Baseline) D-Dimer Inflammatory Biomarker Level
Description: Change from baseline D-Dimer level (Day 1) to maximum level among measures taken during hospitalization and at 30 days. D-Dimer is a small protein fragment present in the blood after a blood clot is degraded by fibrinolysis, so named because it contains two D fragments of the fibrin protein joined by a cross-link.
Time Frame: Baseline (Day 1), Day 30, Days 3 and 7 if hospitalized
Population: Participants with analyzable samples at each timepoint
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Colchicine Plus Current Care | Current Care Alone
Number analyzed (Participants) | 48 | 45
µg/mL
  Baseline: number analyzed (Participants) | 48 | 44
  Baseline | 493.4 (854) | 669 (1101)
  Peak | 638.9 (1112) | 861 (1564)
  Delta: number analyzed (Participants) | 48 | 44
  Delta | 145.5 (353) | 212 (604)

7. Secondary Outcome: Composite Event-Free Survival Over Time (Days)
Description: Participants reaching primary (composite) endpoint were subtracted from event-free survival reported at 10-day intervals
Time Frame: Days 0, 10, 20, 30, 40, 50, 60, 70, 80, and 90
Population: in the rare event of missing data, patients were excluded from analyses
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Plus Current Care | Current Care Alone
Number analyzed (Participants) | 48 | 41
Participants
  Day 0 | 48 | 41
  Day 10 | 40 | 40
  Day 20 | 36 | 38
  Day 30 | 35 | 37
  Day 40 | 35 | 36
  Day 50 | 35 | 36
  Day 60 | 34 | 36
  Day 70 | 34 | 36
  Day 80 | 34 | 36
  Day 90 | 34 | 33

8. Secondary Outcome: Number of Participants Requiring Mechanical Ventilation
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Plus Current Care | Current Care Alone
Number analyzed (Participants) | 48 | 45
Participants | 4 | 2

9. Secondary Outcome: Number of Participants Requiring Mechanical Circulatory Support (MCS)
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Plus Current Care | Current Care Alone
Number analyzed (Participants) | 48 | 45
Participants | 0 | 0

10. Secondary Outcome: Re-hospitalization at 90 Days
Description: Number of participants released and re-admitted to the hospital within 90 days of enrollment
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Plus Current Care | Current Care Alone
Number analyzed (Participants) | 48 | 45
Participants | 7 | 10

11. Secondary Outcome: All-cause Mortality
Time Frame: 90 days
Population: in the rare event of missing data, patients were excluded from analyses
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Plus Current Care | Current Care Alone
Number analyzed (Participants) | 48 | 41
Participants | 8 | 6

ADVERSE EVENTS:
Time Frame: 90 Days
Description: Due to illness of study participants, Adverse Events were recorded as such only if thought to be at least possibly related to study intervention, and not likely due to the primary disease process or its treatment
Arm/Group | Colchicine Plus Current Care | Current Care Alone
All-Cause Mortality (participants affected / at risk) | 8/48 | 6/45
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/45
Other Adverse Events (participants affected / at risk) | 2/48 | 0/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colchicine Plus Current Care (N=48) | Current Care Alone (N=45)
GI discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT04355143/Prot_001.pdf